CLINICAL TRIAL: NCT05846477
Title: Prospective Comparative Monocentric Research Project Study to Compare Cortical Bone Trajectory Screw Insertion Technique With Pedicle Screw Insertion Technique by Use of Patient Specific Drill Guides
Brief Title: MySpine MC Versus MySpine Standard
Acronym: MC vs STD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P05.007.06
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Degenerative Disc Disease; Osteochondrosis; Spondylolysis Lumbar
MeSH Terms: conditions — Intervertebral Disc Degeneration; Osteochondrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- MySpine MC: spinal stabilization via cortical bone trajectory with the support of patient specific guide (MySpine MC technology)
  Interventions: Device: MySpine
- MySpine STD: spinal stabilization via standard pedicle screw positioning with the support of patient specific guide (MySpine std technology)
  Interventions: Device: MySpine

INTERVENTIONS:
Device: MySpine — patient specific guide for screw positioning

SUMMARY:
This research project compares the clinical performance of the cortical bone trajectory CBT insertion technique with the current clinical Gold standard, the Pedicle screw insertion technique. Both techniques are performed by aid of MySpine patient-specific guide systems.

DETAILED DESCRIPTION:
Adult subjects, among those whose clinical condition makes them eligible for a spinal stabilization and meeting the inclusion/exclusion criteria, will be invited to participate to the research project and ask to sign a consent in order to further use of personal and clinical data collected during standard practice visit.

The primary objective of the research project is to compare clinical outcomes, in terms of assessing the main outcomes of importance to patients with back problems (pain, function, symptom-specific well-being, quality of life, disability), of spine surgery with cortical bone trajectory screw placement technique respect the traditional pedicle screw placement technique. Preoperative data and collected during visit as per standard routine at 6 weeks, 3, 6 and 12 months postop will be recoreded and assessed for the purpose of this research project.

ELIGIBILITY:
Inclusion Criteria:

1. patients affected by degenerative disc disease, osteochondrosis and grade I spondylolisthesis needing a one/two level surgical treatment with posterior approach and screw fixation
2. those who need a surgical procedure of lumbar spine stabilization from level L1 to level L5.
3. patients who are willing and able to provide written informed consent for participation in the study. Written informed consent must be obtained prior to the patient's surgery
4. Healthy patients or patients with mild or severe systemic disease identified as patients with ASA score 1, 2 or 3.
5. Patients with BMI ≤ 35 kg/m2
6. non responsive or insufficient response to conservative treatment.

Exclusion Criteria:

1. Patients presenting contraindications as defined by Medacta instruction for use
2. Patients affected by lytic spondylolisthesis and degenerative spondylolisthesis with grade≥2 will be excluded
3. Patients <18 years
4. Patients who are pregnant or intend to become pregnant during the study
5. Known substance or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients listed for lumbar intervertebral body fusion meeting all inclusion/exclusion criteria, will be proposed to take part to the current comparative research project during their pre-operative visit (consecutive ongoing recruitment through project leader in daily clinical practice). They will be provided with an information letter and, in case of acceptance to participate to the research project, asked to sign a consent form in order to further use of personal and clinical data collected during standard practice visit. The patient will be assigned to the research project group according to two consecutive series (First serie: MySpine MC and second serie: MySpine STD).
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Spine surgical patient outcome changing in the time respect the preoperative | baseline, 6 weeks, 3 months, 6 months, 12 months
  Change in Core Outcome Measures Index (COMI) for the assessment of people affected by degenerative lumbar disease in daily practice

SECONDARY OUTCOMES:
Spine Disability index | baseline, 6 weeks, 3 months, 6 months, 12 months
  questionnaire for assessing functional status and quality-of-life impairment in patients with low back pain or spinal cord disease and injury in research and clinical settings.
  he index enquires about functional limitations in various activities of daily living with the index score ranging from 1 (best) to 100 (worst). Among others, pain intensity, personal hygiene, walking, sleeping, social life, sexual life (optional) and travel are assessed by the patient. Each section has six possible responses, which are scored from 0 to 5.
Pain perception | baseline, 6 weeks, 3 months, 6 months, 12 months
  A visual analog scale (from no pain "0" to severe pain "10") to evaluate low back pain
Bone fusion | baseline, 12 months
  A postoperative CT scan will be performed to asses bone fusion at index level defining the presence of bridging bone.
Incidence of adverse event Device-related | baseline, 6 weeks, 3 months, 6 months, 12 months
  Colleciton of all adverse event for all study duration

CONTACTS AND LOCATIONS:
Overall Officials: François Porchet, Dr, Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Switzerland